CLINICAL TRIAL: NCT06431581
Title: Effect of a Mobile Health Intervention on Birth Outcome and Infant Health in a Tertiary Healthcare Facility in Nepal
Brief Title: Effect of a Mobile Health Intervention on Birth Outcome and Infant Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Bhawana Shrestha, Assistant Professor, Kathmandu University School of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NHRC 42-2042
Record Dates: First submitted 2024-05-14; First posted 2024-05-28 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Birth Outcomes; Infant Health
MeSH Terms: interventions — Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (educational video, SMS and reminder phone call) (Experimental): An intervention group will receive standard care along with m-health intervention that includes tailored educational video, SMS and reminder phone call for follow up
  Interventions: Behavioral: m-Health intervention (educational video, SMS and reminder phone call)
- Control Group (standard care, control video and reminder phone call for follow up) (No Intervention): A control group will receive standard care along with a control video and reminder phone call for follow-up

INTERVENTIONS:
Behavioral: m-Health intervention (educational video, SMS and reminder phone call) — Pregnant women meeting the inclusion criteria and assigned to the intervention group will receive m-health intervention that includes a tailored educational video regarding perinatal care targeting positive birth outcomes and infant health, SMS messages, and reminder phone calls for follow-up
  Arms: Intervention group (educational video, SMS and reminder phone call)

SUMMARY:
Globally, neonatal and infant mortality persist as challenging concerns, paralleled by a notable prevalence of low birth weight, preterm birth, and challenges in child growth and development. Some of the factors contributing to these issues include poor maternal health and nutrition, maternal smoking, and insufficient maternal awareness. Despite global efforts to improve maternal, newborn, and child health, adverse birth outcomes remain significant challenges, particularly in low and middle-income countries (LMICs). A noteworthy observation is that not all pregnant women modify their behaviors for their and their baby's health due to lack of social support, fear and insecurity. Recognizing the potential for interventions during pregnancy to positively influence maternal, fetal, and neonatal health, this research underscores the role of Mobile Health (mHealth) technologies in leveraging information and communication technology for health service delivery.

Accordingly, the study aims to evaluate the effect of mobile health intervention on birth outcomes and infant health in Nepal. In the initial phase, a qualitative study will be conducted to explore the enablers and barriers of perinatal care and preferences of pregnant women through focus group discussions. These insights will inform the development of user-centered educational videos and tailored m-Health interventions for pregnant women.

A two-arm parallel randomized controlled trial will then assess the m-Health intervention's effect on the birth outcomes and infant health of the pregnant women attending the antenatal care clinic of Dhulikhel Hospital. The investigaotors will randomize pregnant women at gestational age 14-22 weeks into either a control group (who will receive standard care along with a control video and reminder phone call for follow-up) or an intervention group (who will receive standard care along with m-health intervention that includes educational video, short message service (SMS) and reminder phone call for follow up).

Follow-up will be done from enrollment until the child reaches one year of age, with a focus on evaluating effect of m-Health intervention on birth outcomes (birth weight and gestational age at delivery) and infant health (growth and development of the infant). Data collection will utilize a self-constructed semi-structured questionnaire, along with validated questionnaires. The collected data will be analyzed using STATA 14, contributing valuable insights into the potential effect of m-Health intervention on birth outcomes and infant health.

DETAILED DESCRIPTION:
To evaluate the effect of mobile health intervention on birth outcome and infant health, the sequential exploratory research design will be used. In the initial phase, a qualitative study will be conducted. The researcher and the research assistant will employ purposive sampling to select pregnant women visiting Dhulikhel Hospital in the out patient department (OPD) of the Obstetric department. Written informed consent will be obtained from research participants by either the researcher or research assistant. A focus group discussion will be conducted with pregnant women regarding enablers, barriers, and preferences in perinatal care for improving birth outcomes and infant health. A topic guide will be used for data collection. Subsequently, another focus group discussion will be done with the same participants after developing the educational video to assess the satisfaction and acceptability of the video within the targeted group. The goal of these focus group discussions are to understand the user's needs in educational video. The investigators will ensure that the educational video is user-centered by involving end users (pregnant women) throughout the design and development process. Then after, the content of educational video will be subjected to content validity assessments by subject matter experts to ascertain its accuracy and suitability.

After development and finalization of tailored educational video, a randomized controlled trial will be conducted. Prior to data collection, the researcher will provide information regarding the study such as purpose of the study and assistance required to the health professionals of the antenatal OPD.

Phase 1: Recruitment, baseline data collection and randomization:

The head of the obstetrics and pediatric departments, as well as healthcare professionals at the antenatal care (ANC) clinic and immunization clinic, will be informed about the study. Their active cooperation will be sought throughout the study duration. Pregnant women who are of 14 to 22 weeks of gestation and meet the specified inclusion criteria, while attending the antenatal clinic at Dhulikhel Hospital, will be provided with comprehensive information about the study. This information will cover the study's rationale, procedures, follow-up schedules and voluntary nature of their participation. Eligibility assessments for pregnant women will be conducted by the researcher. Those who expresses a willingness to participate will be asked to provide written informed consent. To ensure impartial allocation of participants to either the intervention or control group, a random sequence number will be generated by a statistician using a computer. These numbers will be securely sealed in envelopes and provided to the enrolled pregnant women. Subsequently, pregnant women who have agreed to participate will be randomized into either the intervention or control group, with a 1:1 ratio, based on the group specified within the sealed envelopes provided to them. The researcher or research assistant will collect baseline information and gather data related to the knowledge of "perinatal care for a healthy birth and a healthy infant" from the participants in both the intervention and control groups.

Phase 2: Delivery of the intervention:

Development of intervention guide: To maintain consistent and standardized delivery of the intervention to all participants, an intervention guide, SMS guide and telephone guide will be developed.

Intervention group: Participants in the intervention group will have access to the educational videos and will be exposed to the following sequence of events:

* During the baseline data collection phase, the initial educational video addressing "perinatal care for a healthy birth and healthy infant" will be viewed by participants via a tablet in a separate designated setting.
* Subsequently, this video will be made available on their smartphones, and participants will be instructed to watch it multiple times during their pregnancy.
* Participants will receive reminder phone calls and SMS to encourage them to watch videos at least three more times after their initial viewing in the antenatal care clinic.
* To ensure continuous engagement, the researcher will maintain regular contact through phone call with intervention group participants, reminding them to view the videos every month from the time of enrollment until delivery and till the child reaches 1 year of age as per the reminder schedule.
* Additionally, pregnant mothers will be explicitly instructed to discuss the video content solely with their immediate family members and refrain from sharing it with others.

Control group: In contrast, participants in the control group will receive usual standard care and will be allowed to view a control video. Participants will be contacted through phone calls to remind their follow-up visit.

Phase 3: Follow up

Participant assessment and follow-up: The participants from both the intervention and control groups will undergo a series of assessments and follow -up visits.

• Post intervention knowledge assessment: Following the intervention phase, both groups will be subjected to a post-intervention knowledge assessment. The overall knowledge of perinatal care for birth outcome and infant health will be assessed approximately one month following the participants' initial viewing of the videos.

• Birth outcome assessment: Both the intervention and control group participants will be followed up within the first 24 hours of their delivery to evaluate and record the birth outcomes.

• Infant health assessment: In the subsequent phase of the study, which aims to evaluate the impact of the intervention on infant health, the growth and development of infant will be assessed. Both groups will be informed of the necessity of follow-up visits at the immunization clinic through phone calls. Following the notification, the growth and developmental assessments of the infants will be conducted at the immunization clinic on the day of their scheduled immunization visit (at 6 weeks, 14 weeks, 9 months, and 12 months of life). For those participants who are unable to visit immunization clinic of Dhulikhel Hospital, they will be followed up at their nearby health post or within their homes. This follow-up process will be conducted by the researcher, along with the assistance of a research assistant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of age 18 years and above;
* Pregnant with 14 to 22 weeks of gestation;
* Planned to deliver a child and come for infant's vaccination at Dhulikhel hospital;
* Pregnant women who use smart phone;
* Pregnant women who have plan to stay in Dhulikhel thorough out this study period;
* Can read and understand Nepali language

Exclusion Criteria:

* Vision impairment and diagnosed learning difficulties

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Birth weight | 1-1.5 years
  The birth weight of the newborns delivered from the participants will be measured in grams. The mean birth weight of the newborns in both the intervention group and the control group will be compared.
Gestational age at delivery | 1-1.5 years
  The gestational age at delivery will be expressed in completed weeks of gestation. The mean gestational age at delivery will be compared between the intervention group and the control group.

SECONDARY OUTCOMES:
Knowledge on perinatal care | 6 months
  Knowledge on perinatal care for healthy birth and healthy infant will be assessed through validated knowledge related questionnaire. The mean score will be be calculated for both the intervention and the control group and then will be compared.
Weight of the infant | 2-2.5 years
  The weight of the infant will be measured in grams and compared to the World Health Organization(WHO) standard for weight-for-age of the infant.
Height/Length of the infant | 2-2.5 years
  The height/length of the infant will be measured in centimeters and compared to the WHO standard for height-for-age of the infant.
Development of an infant | 2-2.5 years
  The development of an infant will be evaluated using the Ages and Stages Questionnaire (ASQ) and average ASQ score will be determined

CONTACTS AND LOCATIONS:
Locations (1):
- Bhawana Shrestha, Dhulikhel, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lassi ZS, Middleton PF, Crowther C, Bhutta ZA. Interventions to Improve Neonatal Health and Later Survival: An Overview of Systematic Reviews. EBioMedicine. 2015 May 31;2(8):985-1000. doi: 10.1016/j.ebiom.2015.05.023. eCollection 2015 Aug. PMID 26425706
- [Background] Khani Jeihooni A, Mohammadkhah F, Razmjouie F, Harsini PA, Sedghi Jahromi F. Effect of educational intervention based on health belief model on mothers monitoring growth of 6-12 months child with growth disorders. BMC Pediatr. 2022 Sep 23;22(1):561. doi: 10.1186/s12887-022-03593-8. PMID 36151526
- [Background] Lassi ZS, Mansoor T, Salam RA, Das JK, Bhutta ZA. Essential pre-pregnancy and pregnancy interventions for improved maternal, newborn and child health. Reprod Health. 2014;11 Suppl 1(Suppl 1):S2. doi: 10.1186/1742-4755-11-S1-S2. Epub 2014 Aug 21. PMID 25178042
- [Background] Taneja S, Chowdhury R, Dhabhai N, Mazumder S, Upadhyay RP, Sharma S, Dewan R, Mittal P, Chellani H, Bahl R, Bhan MK, Bhandari N; Women and Infants Integrated Growth Study (WINGS) Group. Impact of an integrated nutrition, health, water sanitation and hygiene, psychosocial care and support intervention package delivered during the pre- and peri-conception period and/or during pregnancy and early childhood on linear growth of infants in the first two years of life, birth outcomes and nutritional status of mothers: study protocol of a factorial, individually randomized controlled trial in India. Trials. 2020 Jan 31;21(1):127. doi: 10.1186/s13063-020-4059-z. PMID 32005294
- [Background] Toolan M, Barnard K, Lynch M, Maharjan N, Thapa M, Rai N, Lavender T, Larkin M, Caldwell DM, Burden C, Manandhar DS, Merriel A. A systematic review and narrative synthesis of antenatal interventions to improve maternal and neonatal health in Nepal. AJOG Glob Rep. 2022 Feb;2(1):100019. doi: 10.1016/j.xagr.2021.100019. PMID 35252905
- [Background] Park JJH, Harari O, Siden E, Zoratti M, Dron L, Zannat NE, Lester RT, Thorlund K, Mills EJ. Interventions to improve birth outcomes of pregnant women living in low- and middle-income countries: a systematic review and network meta-analysis. Gates Open Res. 2020 Sep 24;3:1657. doi: 10.12688/gatesopenres.13081.2. eCollection 2019. PMID 33134854
- See also: Effect of parenting intervention through "Care for Child Development Guideline" on early child development and behaviors: a randomized controlled trial. BMC Pediatr.2022;22(1):690 — https://doi.org/10.1186/s12887-022-03752-x
- See also: Pregnancy and Childbirth - Healthy People 2030 | health.gov — https://health.gov/healthypeople/objectives-and-data/browse-objectives/pregnancy-and-childbirth
- See also: Lessons from digital technology-enabled health interventions implemented during the coronavirus pandemic to improve maternal and birth outcomes: a global scoping review. BMC Pregnancy Childbirth. 2023 Mar 20;23(1):195. — https://doi.org/10.1186/s12884-023-05454-3